CLINICAL TRIAL: NCT04841239
Title: Development of Topical Herbal Formulations for Treatment of Cutaneous Leishmaniasis: A Single Blind, Randomized, Placebo Controlled Preclinical and Clinical Trials
Brief Title: Development of Topical Herbal Formulations for Treatment of Cutaneous Leishmaniasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jinnah Sindh Medical University (Other)
Responsible Party: Principal Investigator, Muhammad Arif Asghar, Principal Investigator, Jinnah Sindh Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DISDSK-937/-22
Record Dates: First submitted 2021-04-05; First posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Leishmaniasis, Cutaneous
MeSH Terms: conditions — Leishmaniasis, Cutaneous

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Herbal topical formulation (Experimental)
  Interventions: Other: Herbal topical formulation
- Control (No Intervention)

INTERVENTIONS:
Other: Herbal topical formulation
  Arms: Herbal topical formulation

SUMMARY:
Infections due to protozoa of the genus Leishmania are a major worldwide skin problem, with high endemicity in developing countries including Pakistan. As far as concern for the treatment of cutaneous leishmaniasis (CL), there is no single therapeutic agent that has proved a satisfactory efficacy and safety. Therefore, the objective of this research study was to develop an alternative therapeutic approach for the treatment of CL. In the current research protocol, two herbal topical formulations (Gyburene and Thuscare) were prepared containing to contain 5% Casuarina equisetifolia L. and Thespesia populnea L. plant extract and evaluate their leishmanicidal potential in pre-clinical and randomized clinical trials studies. Preclinical studies were performed on BALB/c mice after the development of a lesion on the dermis caused by the Leishmania (L.) major parasite. Six weeks randomized, single single-blind placebo controlled study was also conducted on seventy eight L. major infected patients divided into three groups i.e. treated, reference and placebo with the 1:1 ratios.

DETAILED DESCRIPTION:
STUDY PROTOCOL

1.1. Introduction Leishmaniasis is a major neglected health problem frequently found in tropical and subtropical regions with the prevalence rate of 1.5 million per year globally. The disease is caused by protozoan parasite from genus Leishmania. Transmission occurred by sand fly of genus Phlebotomus in the (Old World) and Lutzomyia (New World). Cutaneous leishmaniasis is restricted to skin and around 185 million people at risk in 61 countries. Now it is endemic in Pakistan (different regions) and diffuses fastly, particularly in the refugee camps main causative agent found is L. major followed by L. tropica. Vigilant literature review revealed that besides the four provinces of Pakistan increased incidences of CL were found in Balochistan which is largest province (in area) followed by NWFP. In Sindh province (Dadu, Jacobabad, Larkana and Karachi) are commonly reported for cases while in Punjab (Multan and Dera Ghazi Khan) are mainly reported for the occurrence of disease. Diagnosis of this diseases is done by clinical picture usually dry lesions are caused by L. tropica while moist and early ulcerative lesions are caused by L. major, such lesions take months to years for healing eventually heal by own but satellite lesions and bacterial and fungal infections results in delayed and complicated healing process, but in non-endemic areas it is difficult to diagnose because of unclear form, along with this secondary infections, delay treatment as well as mistreatment sometimes can also cause changes in clinical picture. In such situations examination of smear from lesion is the diagnostic tool along with culture and histopathological examinations.

1.2. Clinical trials against CL Methanolic bark extract of Casuarina equisetifolia L. showed good antileishmanial potential against L.major using in vitro analysis which directed us towards an innovative therapeutic concept for development of new herbal formulations against leishmaniasis through accelerated wound closures in clinical trials on human contestants. Ulcerative CL is because of defective wound healing depending on this hypothesis current study is planned to explored clinical efficacy of new protocol Gyburene 5% cream as anti-parasitic agent followed by Thuscare 5% ointment for speed up wounds closure. The primary objective of this study is to evaluate anti leishmanial outcome of Gyburene 5% cream at wound closure and after six months while secondary objective is to evaluate that incessant wound care along with anti-parasitic agent can results in valuable enhancement in treatment.

1.3. Sample population and study design: This is a single-blind, randomized study. Seventy patients with confirmed with cutaneous leishmaniasis were recruited in the study. Participants were randomly allocated into two groups. Pilot group (did not receive any medication before) and resistant group (who already received medication either parental or topical). During trials 20 participants were dropped as a result of lack of follow up specially the affected people coming from rural areas.

1.3.1. Ethical consideration: The research protocol was approved by ethical committee of the Board of Advanced Studies and Research University of Karachi Vide Resol No. 16. Informed consents forms were taken from each patient.

1.3.2. Patient Assessment:

Medical history of each patient (age, sex, co-morbidities, wound condition, site and size of lesion with Giemsa smear test report) was taken prior to treatment protocol on clinical Performa specially designed for this study and consisted of two parts, first for personnel information and second for medical history. Lesion size was calculated using Vernier caliper in two dimensions and each participant advised for weekly follow up till end of therapy, portrait photograph were taken before, throughout and after therapy using digital camera for assessment of healing percentage. Cured patients follow up was done for further six months to ensure no set back has been happened. Presence or absence of parasite was confirmed by smear test while healed area was calculated by percentage of healing by following formula (Baie and Sheikh, 2000):

1.3.2.1. Inclusion criteria

1. Patients who met the histological criteria for presence of parasite
2. Age of older than 4 years and both gender.
3. Lesions are less than 5 in number in each patient
4. Size of lesion is less than 5cm2
5. Participants who had stopped therapy greater than 4 weeks earlier and the lesions were not improving.
6. Duration of disease for patients under trial was six months (acute) and more than one year (chronic).

1.3.2.2. Exclusion criteria

1. Patients who had taken any immuosuppressive drugs or anti leishmanial drugs in last month.
2. Pregnant women and lactating mothers.
3. Contestants with complications of renal, hepatic and pulmonary disease, Immune-o- compromised patients such as (HIV).
4. Patients suffering from conditions like malaria, tuberculosis and treatment regimen is going on for such infections.

1.3.3. Study treatment Prior to the initiate treatment protocol toxicological evaluation of herbal extracts was also done to ensure the safety of topical herbal pharmaceutical preparations. In case of more than one lesion any one targeted for biopsies although all received same treatment. Both groups of patient were treated with topical herbal formulations Gyburene 5% cream (for cure of CL) in morning and evening and Thuscare 5% ointment (for rapid wound healing and cure of super infections) only at night in two different directions at the angle of 90º to each other by leaving lesion uncovered.

Before application of second formulation all contestant were advised to wash the lesion with normal saline. Weekly follow up was done till completion of the therapy in order to ensure the entire cure such as for negative smear skin test amastigotes in Giemsa strain and complete healing with re-epithelialization of the lesion. Each formulation was dispensed in 10 g container (separately) enough for one week.

1.4. Statistical Analysis T-test used for comparison rate of healing between two groups while Kaplan Meier test between pilot and resistant group while Kaplan Meier test used to calculate healed area per week for both resistant and pilot group at P<0.05 using SPSS version 21.

Clinical evaluation Performa for Cutaneous Leishmaniasis (CL) Personal information Patient code: ------------------- Male/Female: ---------------------- Age: ---------- Address: --------------- Occupation: ------------------- Marital status: -------------

Contact No: -------------------------- CNIC No: ------------------------Family history:

Clinical information Morphology of lesion

* Ulcerated
* Crust
* Plaque
* Nodule Lesion condition
* Dry
* Wet Giemsa Smear test
* Positive
* Negative Duration of lesions
* ≥ 6 month
* Between 6-12 months
* ≤ 6 month No of lesions
* 1
* 2
* 3
* 4
* 5

Health condition

* Arthritis
* Allergy
* Diabetes
* Immune disorder
* Blood pressure Differential diagnosis for CL
* Bacterial and fungal skin infection
* Eczema
* Syphilis
* Sarcoidosis
* Blastomycosis
* Others Area of lesion/visit Visit I: Area=……………cm2 Visit II: Area= …………..cm2 Visit III: Area=…………. cm2 Visit IV: Area=………… cm2 Visit V: Area=…………. cm2

Remarks of Dermatologist:

Signature of Dermatologist

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for participants including;

  * • Patients who met the histological criteria for presence of parasite
  * Age of older than 4 years and both gender.
  * Lesions are less than 5 in number in each patient
  * Size of lesion is less than 5cm2
  * Participants who had stopped therapy greater than 4 weeks earlier and the lesions were not improving.
  * Duration of disease for patients under trial was six months (acute) and more than one year (chronic).

Exclusion Criteria:

* The following patients were excluded:

  * Whose clinical data were incomplete
  * Participants who had received any anti anti-leishmanial or immunosuppressive drugs in the last 15 days
  * Patients with co-morbid conditions, immunocompromised patients,
  * Lactating mothers and pregnant women.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2014-12-30 (Actual); Study Completion 2014-12-30 (Actual)

PRIMARY OUTCOMES:
The lesion progression was followed microscopically and the strain presence present in biopsy material was also confirmed microscopically in both cultures and smears after six weeks treatment. | 6 weeks
  The primary endpoint of leishmaniasis cure from topical herbal formulations was assessed microscopically in both cultures and smears.

SECONDARY OUTCOMES:
Measurement of lesions size between placebo, treated and reference groups after the six weeks treatment period | 6 weeks
  For the monitoring of healing progressed, photographs were taken before, during and after completion of therapy using a digital camera while healed area was calculated by percentage of healing by following formula:
  Healed area percent of wound contraction = ………………………………. ×100 Total area before treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yousra Shafiq, Ph.D, Principal Investigator — Jinnah Sindh Medical University
Locations (1):
- Civil Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
All types of data after publication on request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After study will be published
Access Criteria: On request